CLINICAL TRIAL: NCT01175057
Title: Pilot Study for Evaluation of the MeDiNa Concept of Homely Rehabilitation of Patients With Acute Myocardial Infarction
Brief Title: MeDiNa Pilot Study for Evaluation of the MeDiNa Concept of Homely Rehabilitation After Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Collaborators: Philips Healthcare (Industry); MUL Services GmbH (Unknown); Fraunhofer Institute (IMS) (Unknown)
Responsible Party: Sponsor
Other Study IDs: Medina Pilot Study
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Feasibility of Telemedical Home Monitoring; Post Stationary; Patients With Myocardial Infarction
Keywords: feasibility; compliance; telemedical home monitoring; post stationary rehabilitation; patients with myocardial infarction
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: 10 patients who undergo home monitoring with the MeDiNa Homebox for 4 weeks and then 4 weeks without the MeDina Homebox
- Group B: Group B starts without the MeDiNa Homebox for 4 weeks and then undergo Homemonitoring with the MeDiNa Homebox for 4 weeks.

SUMMARY:
In this study feasibility of the MeDiNa concept is looked at, which means telemedical services for homely rehabilitation. With the help of microsystems technology, the relevant vital signs are measured at the patient's home, then transmitted to the MeDiNa- Homebox- Tablet PC (by bluetooth) and then transferred into a central database, the MeDiNa eHealth- portal (by HSDPA, UMTS). These parameters can be continuously monitored by authorized network participants such as the family doctor or the patients themselves. In future, beyond cost advantages this will help to supervise risk patients or inspire patients to take more care of their health during homely rehab.

DETAILED DESCRIPTION:
Patients after myocard infarction who undergo homely rehab post stationary are divided into two groups of 10 patients each. The patients of group A undergo home monitoring for 4 weeks with the MeDiNa Homebox and afterwards 4 weeks without home monitoring. Group B starts vice versa, without home monitoring first and then undergoes home monitoring for 4 weeks (cross over,controlled intra-individually). During home monitoring with the MeDiNa Homebox patients measure vital parameters (weight, blood pressure, ECG (by chest strap including micro sensors), pulse and activity (also by chest strap including accelerometer) several times a day. The pseudonomized data which are transferred via the MeDiNa Homebox- Tablet PC to the MeDiNa eHealth Internet Portal (UMTS, HSDPA) to which the responsible authorized medicines will have access will be evaluated descriptively.

ELIGIBILITY:
Inclusion Criteria:

* female and male patients minimum 60 years old
* myocardial infarction
* post stationary rehabilitation at home
* Internet access or mobile phone reception possible
* able to give informed consent

Exclusion Criteria:

* patients with dementia
* aphasic impairment
* serious pulmonary diseases
* motional resriction (e.g. amputee)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Medical Clinic I, RWTH Aachen University Hospital, Pauwelsstaße 30, 52074 Aachen, post stationary after myocardial infarction and who are at least 60 years old
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of feasibility of telemedical home monitoring with the MeDiNa concept with patients after myocard infarction post stationary who undergo homely rehab | 8 weeks for each patient, about 6 months totally
  Patients are divided into two groups of 10 patients.The patients of group A undergo home monitoring for 4 weeks with the MeDiNa Homebox and afterwards 4 weeks without home monitoring. Group B starts vice versa (cross over, controlled intra-individually). During home monitoring with the MeDiNa Homebox patients measure vital parameters (weight, blood pressure, pulse, ECG) several times a day. The data are sent to the MeDiNa Homebox (by Bluetooth) and then to an Internet Portal (by USMB, HSDPA), to which the responsible authorized medicine will have access.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Krüger, PD Dr. med., Principal Investigator — RWTH Aachen University, Department of Cardiology, Pulmonology and Vascular Medecine Aachen, NRW, Germany
Locations (1):
- Medical Clinic I, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany